CLINICAL TRIAL: NCT00646477
Title: Therapeutic Efficacy Evaluation of the CPAP/autoCPAP Sandman in the Treatment of New Patients With Obstructive Sleep Apnoea Syndrome
Brief Title: ISIS 1 Therapeutic Effectiveness
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tyco Healthcare Group (Industry)
Responsible Party: EMEA Clinical Affairs - Respiratory & Monitoring Solutions, Tyco Healthcare Group
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 1
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: OSAS (Obstructive Sleep Apneas Syndrome)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): Phase 1 : manual Phase 2 : automatic Descent rate pressure : slow
  Interventions: Device: titration night
- B (Experimental): Phase 1 : manual Phase 2 : automatic Descent Rate Pressure : fast
  Interventions: Device: titration night
- C (Experimental): Phase 1 : automatic Phase 2 : manual Descent rate pressure : slow
  Interventions: Device: titration night
- D (Experimental): Phase 1 : automatic Phase 2 : manual Descent Rate Pressure : fast
  Interventions: Device: titration night

INTERVENTIONS:
Device: titration night — Each subject undergo 1 night of full polysomnography split into 2 consecutives and randomized sequences, using the Sandman device into two different modes:
  in APAP mode - Data analysis of this sequence will be used to evaluate the therapeutic effectiveness of the CPAP/autoCPAP Sandman in APAP mode compared both to the polysomnography registration and the diagnosis night for each enrolled patient. The type of respiratory events and their index/hour of sleep and the total arousal index will be appraised as markers of the efficacy of OSAS treatment, constituting the primary outcomes.
  in CPAP mode for manual titration sequence.During the manual titration, 5 constant pressure levels settings were studied for equal periods of 30 minutes gradually increasing the pressure. The aim of this sequence is to determine the sensitivity and the specificity of the CPAP/autoCPAP Sandman in detecting respiratory events.

SUMMARY:
The study is a prospective field evaluation to assess the therapeutic value of the CPAP/autoCPAP Sandman in 24 new diagnosed Obstructive Sleep Apneic patients.

Precisely, the study was designed to :

* evaluate the therapeutic efficacy of the CPAP/autoCPAP Sandman device in improving sleep quality and normalozing respiratory events
* determine the sensitivity and specificity of the device in adequately detecting respiratroy events
* compare effective pressure Peff determined by the device and during manual titration
* compare the impact of the two-speed descent pressure algorithm

DETAILED DESCRIPTION:
During the study, each patient underwent one night of full polysomnography with two consecutives therapeutic sequences during the same night, after randomization of the passage order:

* autotitrating pressure phase: sleep parameters and respiratory events vs results of the polysomnographic registration,
* manual titration phase: concordance between events respiratory analyzed on the polysomnographic recordings and the events detected by the CPAP / auto-CPAP.

ELIGIBILITY:
Inclusion Criteria:

* patient male or female, aged 18 to 75 years
* weight > 30kg
* patient with a newly diagnosed OSAS, under treatment with CPAP
* patient in stable condition
* patient affiliated to a social security insurance
* having given its written informed consent to participate to the study

Exclusion Criteria:

* pneumothorax or pneumomediastin history
* massive epistaxis (current or previous)
* decompensated heart failure or hypotension
* pneumoencephal history, recent trauma or surgery sequel with cranio-nasopharyngeal fistula
* acute sinusitis history, middle ear infection or perforation of the tympanic membrane
* respiratory insufficiency or severe respiratory illness with the possibility of residual hypoxemia
* severe bullous emphysema or previously complicated pneumothorax
* severe claustrophobia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
To determine the sensitivity and specificity of the CPAP/autoCPAP Sandman in adequately detecting respiratory events and to evaluate the therapeutic effectiveness of the device in improving sleep quality and normalizing respiratory events | May 2008

SECONDARY OUTCOMES:
To compare effective pressure Peff determined by the device and during manual titration | May 2008
To compare the impact of the two-speed descent pressure algorithm | May 2008

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Grillier-Lanoir, Study Chair — Tyco Healthcare Group
Locations (1):
- Hospital Michalon, sleep disorders center, Grenoble, France